CLINICAL TRIAL: NCT01024075
Title: The Adjunctive Use of a Dexamethasone-Sinufoam Mixture on Endoscopic Sinus Surgery Outcomes: A Randomized, Double-Blind, Placebo-controlled Trial
Brief Title: Effect of Sinufoam-Dexamethasone Mixture on Post Endoscopic Sinus Surgery Outcomes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Luke Rudmik, MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22476
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic Rhinosinusitis; Endoscopic sinus surgery; Sinufoam; Dexamethasone; For patients with Chronic Rhinosinusitis without nasal polyps; Focus: Define the postoperative sinonasal mucosal healing status of 2 Sinufoam mixtures
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Sinufoam is mixed with saline and placed within the ethmoid cavity at the completion of sinus surgery
  Interventions: Drug: Saline
- Dexamethasone (Active Comparator): Sinufoam is mixed with dexamethasone and placed within the ethmoid cavity at the completion of sinus surgery
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 4cc of Dexamethasone and 4cc of Saline mixed with Sinufoam
  Arms: Dexamethasone
Drug: Saline — 8cc of Saline mixed with Sinufoam
  Arms: Saline

SUMMARY:
Dexamethasone added to sinufoam, which is placed in the ethmoid cavity at the completion of endoscopic sinus surgery, will improve sinonasal mucosal healing.

DETAILED DESCRIPTION:
Sinufoam is an FDA approved mixture, which is placed in the ethmoid cavity at the completion of an endoscopic sinus surgery procedure. Sinufoam prevents scarring and promotes healing of the sinonasal mucosa. Sinufoam is commonly mixed with saline, which enables it to be liquefied and gently placed into the ethmoid cavity. Recent practice of adding Dexamethasone to the sinufoam mixture has been hypothesized to promote healing by reducing chronic inflammation associated with CRS. Using topical dexamethasone mixed into the Sinufoam solution may improve patient care by preventing the systemic effects associated with post-operative systemic steroid use.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Chronic Rhinosinusitis without nasal polyps --- defined according to the AAO guidelines
* Elective "Bilateral" sinus surgery requiring at a minimum of an Uncinectomy, Maxillary Antrostomy, and Anterior Ethmoidectomy.

Exclusion Criteria:

* Uncorrectable coagulopathy
* Emergency procedure
* Unavailable for standard post operative follow-up
* Sinonasal neoplasm resections
* Excessive intra-operative bleeding requiring nasal packing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Sinonasal mucosal healing | 1 month

SECONDARY OUTCOMES:
Sinonasal quality of life (SNOT-22) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Luke Rudmik, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Rudmik L, Mace J, Mechor B. Effect of a dexamethasone Sinu-Foam middle meatal spacer on endoscopic sinus surgery outcomes: a randomized, double-blind, placebo-controlled trial. Int Forum Allergy Rhinol. 2012 May-Jun;2(3):248-51. doi: 10.1002/alr.21011. Epub 2012 Jan 17. PMID 22253199